CLINICAL TRIAL: NCT02992496
Title: Investigation of Antidepressant Efficacy of Oral Ketamine Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Assoc.-Prof., MD PD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: v1.2_20161024
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Major Depressive Episode
MeSH Terms: interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine treatment group (Active Comparator): Each patient will undergo six treatment sessions with 1mg/kg oral ketamine over 2 weeks.
  Interventions: Drug: Ketamine
- Control group (Active Comparator): Each patient will undergo six treatment sessions with 0.03mg/kg oral midazolam over 2 weeks
  Interventions: Drug: Midazolam Hydrochloride

INTERVENTIONS:
Drug: Ketamine — 1mg/kg, 6 applications over 2 weeks
  Arms: Ketamine treatment group
Drug: Midazolam Hydrochloride — 0.03mg/kg, 6 applications over 2 weeks
  Arms: Control group

SUMMARY:
The purpose of this double-blind, controlled, randomized study is to investigate the antidepressant efficacy of oral ketamine treatment in patients suffering from a major depressive episode.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a major depressive episode in the scope of a major depressive or bipolar disorder supported by a Structured Clinical Interview for DSM-IV-TR (SCID)
* Hamilton depression rating scale score ≥ 19
* Willingness and competence to sign the informed consent form
* Stable psychopharmacological treatment for 10 days (except benzodiazepines)

Exclusion Criteria:

* Initiation of a new antidepressant or mood stabilizing treatment (pharmacological, physical or psychotherapeutic) with adequate dosage (as defined by the minimum recommended dose in the respective prescribing information) within 4 weeks prior to inclusion
* Prior use of ketamine
* Pregnancy/Breast feeding
* Instable arterial hypertension >170/110mmHg
* Hepatic dysfunction
* Hyperthyreosis
* History of glaucoma
* Neurodegenerative disorders
* Any unstable medical illness
* History of substance abuse within the past 12 months
* History of psychosis
* Failure to comply with the study protocol or to follow the instructions of the investigating team
* Current treatment with one of the following drugs: clopidogrel, carbamazepine, valproate, barbiturates, memantine, modafinil, disulfiram, amiodarone, ranolazine, phenytoin, verapamil, fibrates, antiretroviral agents, antimicrobial chemotherapeutics, azole antifungals, glucocorticoids, cyclosporine, valeriana/garlic/grapefruit preparations, St. John's wort.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 1 week

SECONDARY OUTCOMES:
Clinician Administered Dissociative States Scale (CADSS) | 2 weeks
Hamilton Depression Rating Scale | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No